CLINICAL TRIAL: NCT07255729
Title: Machine Learning-Based Exosomal microRNA Signature for Preoperative Staging and Chemotherapy Eligibility in Colon Cancer
Brief Title: An Exosomal microRNA Signature for Preoperative Staging in Colon Cancer
Acronym: EXPOSE
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/EXPOSE
Record Dates: First submitted 2025-11-17; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Colon Cancer
Keywords: CC; NAC; miRNA; Exosomal miRNA; Staging; liquid biopsy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma or serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- High-risk Colon Cancer (Discovery): Stage IIB-IV colon cancer; used to identify biomarker candidates
  Interventions: Diagnostic Test: Diagnostic Test: EXPOSE assay（Small RNA-seq of exosomal miRNAs）
- Low-risk Colon Cancer (Discovery): Stage I-IIA colon cancer
  Interventions: Diagnostic Test: Diagnostic Test: EXPOSE assay（Small RNA-seq of exosomal miRNAs）
- High-risk Colon Cancer (Training): Pathological Stage IIB-IV; used to build model
  Interventions: Diagnostic Test: Diagnostic Test: EXPOSE RT-qPCR panel
- Low-risk Colon Cancer (Training): Pathological Stage I-IIA
  Interventions: Diagnostic Test: Diagnostic Test: EXPOSE RT-qPCR panel
- High-risk Colon Cancer (Validation): Stage IIB-IV in independent cohort
  Interventions: Diagnostic Test: Diagnostic Test: EXPOSE RT-qPCR panel
- Low-risk Colon Cancer (Validation): Stage I-IIA in independent cohort
  Interventions: Diagnostic Test: Diagnostic Test: EXPOSE RT-qPCR panel

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: EXPOSE assay（Small RNA-seq of exosomal miRNAs） — Candidates identified from small RNA sequencing
  Groups: High-risk Colon Cancer (Discovery); Low-risk Colon Cancer (Discovery)
Diagnostic Test: Diagnostic Test: EXPOSE RT-qPCR panel — Quantification of exosomal microRNAs (RT-qPCR)
  Groups: High-risk Colon Cancer (Training); High-risk Colon Cancer (Validation); Low-risk Colon Cancer (Training); Low-risk Colon Cancer (Validation)

SUMMARY:
Recent studies have highlighted the potential benefits of neoadjuvant chemotherapy (NAC) in colon cancer; however, its indication is generally limited to cases corresponding to pathological stage IIB or higher. Accurately identifying such high-risk cases before surgery remains challenging using conventional clinical diagnostics alone. Therefore, we hypothesized that integrating molecular biomarkers with preoperative clinical assessment could provide a more precise and sensitive evaluation of tumor aggressiveness. In this context, we focused on exosomal microRNAs, which are actively secreted from tumor cells and remain stable in circulation, and aimed to develop a machine learning-based biomarker panel. To achieve this, we initiated a multicenter study utilizing preoperative plasma samples to establish a reliable biomarker model for risk stratification and treatment decision-making in colon cancer.

DETAILED DESCRIPTION:
Colon cancer remains one of the leading causes of cancer-related mortality worldwide, and despite advances in screening and surgical techniques, a substantial proportion of patients continue to experience disease recurrence after curative resection. For patients with pathological stage IIB or higher disease, adjuvant chemotherapy is routinely recommended due to their elevated recurrence risk. However, accurately identifying these biologically aggressive cases before surgery remains a major clinical challenge, as current imaging-based staging often underestimates tumor burden and fails to capture underlying malignant potential. This diagnostic gap has hindered the optimal implementation of neoadjuvant chemotherapy (NAC) in colon cancer.

To address this issue, the investigators established the EXPOSE study (Exosomal microRNA Signature for Pre-Operative Stage and Eligibility Evaluation), a multicenter translational research initiative aiming to develop and validate a noninvasive, biologically informed diagnostic assay capable of identifying patients with high-risk colon cancer-equivalent to pathological stage IIB or higher-who may benefit from NAC.

The EXPOSE study will proceed through three structured phases.

1. In the discovery phase, exosomal microRNAs will be profiled using comprehensive small RNA sequencing to identify key biomarkers reflecting tumor aggressiveness.
2. In the training phase, the investigators will quantify candidate microRNAs using RT-qPCR and integrate their expression patterns via machine-learning algorithms to construct a predictive model for high-risk disease.
3. Finally, in the validation phase, the model's reproducibility, diagnostic accuracy, and generalizability will be tested in an independent clinical cohort.

The final EXPOSE assay is expected to serve as a liquid biopsy-based tool for preoperative staging, enabling more precise identification of biologically advanced colon cancer cases. Upon completion, this study will deliver a rigorously validated diagnostic model that combines molecular and clinical data to guide neoadjuvant treatment decisions and enhance personalized care in colon cancer management.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed colon cancer (Stage I-IV, UICC TNM 8th edition)
* Underwent curative-intent resection (with or without perioperative therapy)
* Preoperative plasma (or serum) samples available
* Clinical and prognostic data available

Exclusion Criteria:

* No written informed consent
* Missing preoperative blood samples
* Missing survival/recurrence data
* Duplicate cases
* Non-adenocarcinoma histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon cancer patients (Stage I-IV) from multiple institutions with preoperative serum or plasma samples and complete pathological staging.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Pathological Stage IIB or higher patients | At time of pathology (1year after surgery)

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 120 months
Overall survival (OS) | Up to 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Morgan E, Arnold M, Gini A, Lorenzoni V, Cabasag CJ, Laversanne M, Vignat J, Ferlay J, Murphy N, Bray F. Global burden of colorectal cancer in 2020 and 2040: incidence and mortality estimates from GLOBOCAN. Gut. 2023 Feb;72(2):338-344. doi: 10.1136/gutjnl-2022-327736. Epub 2022 Sep 8. PMID 36604116
- [Background] Cardoso R, Guo F, Heisser T, Hackl M, Ihle P, De Schutter H, Van Damme N, Valerianova Z, Atanasov T, Majek O, Muzik J, Nilbert MC, Tybjerg AJ, Innos K, Magi M, Malila N, Bouvier AM, Bouvier V, Launoy G, Woronoff AS, Cariou M, Robaszkiewicz M, Delafosse P, Poncet F, Katalinic A, Walsh PM, Senore C, Rosso S, Vincerzevskiene I, Lemmens VEPP, Elferink MAG, Johannesen TB, Korner H, Pfeffer F, Bento MJ, Rodrigues J, Alves da Costa F, Miranda A, Zadnik V, Zagar T, Lopez de Munain Marques A, Marcos-Gragera R, Puigdemont M, Galceran J, Carulla M, Chirlaque MD, Ballesta M, Sundquist K, Sundquist J, Weber M, Jordan A, Herrmann C, Mousavi M, Ryzhov A, Hoffmeister M, Brenner H. Colorectal cancer incidence, mortality, and stage distribution in European countries in the colorectal cancer screening era: an international population-based study. Lancet Oncol. 2021 Jul;22(7):1002-1013. doi: 10.1016/S1470-2045(21)00199-6. Epub 2021 May 25. PMID 34048685
- [Background] Taieb J, Svrcek M, Cohen R, Basile D, Tougeron D, Phelip JM. Deficient mismatch repair/microsatellite unstable colorectal cancer: Diagnosis, prognosis and treatment. Eur J Cancer. 2022 Nov;175:136-157. doi: 10.1016/j.ejca.2022.07.020. Epub 2022 Sep 14. PMID 36115290
- [Background] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766
- [Background] Burley N, Lee Y, Liu L, Gangi A, Nasseri Y, Atkins K, Zaghiyan K, Murrell Z, Osipov A, Hendifar A, Hitchins M, Gong J. ctDNA-guided adjuvant immunotherapy in colorectal cancer. Immunotherapy. 2024;16(20-22):1197-1202. doi: 10.1080/1750743X.2024.2430941. Epub 2024 Nov 17. PMID 39552190
- [Background] Tan PB, Verschoor YL, van den Berg JG, Balduzzi S, Kok NFM, Ijsselsteijn ME, Moore K, Jurdi A, Tin A, Kaptein P, van Leerdam ME, Haanen JBAG, Voest EE, de Miranda NFCC, Schumacher TN, Wessels LFA, Chalabi M. Neoadjuvant immunotherapy in mismatch-repair-proficient colon cancers. Nature. 2025 Dec;648(8094):726-735. doi: 10.1038/s41586-025-09679-4. Epub 2025 Oct 20. PMID 41115454
- [Background] Krsul D, Prenc E, Pozgaj L, Stefok D, Pongrac P, Podolski M, Radicevic AP, Karlovic D, Jerkovic A, Golcic M, Drazic I, Glavas Krsul S, Fuckar Cupic D, Erakovic Haber V, Zelic M. Diagnostic Relevance of miR-185, miR-141, and miR-21 in Colon Carcinoma: Insights into Tumor Sidedness and Reference Gene Selection. Biomedicines. 2025 Oct 10;13(10):2460. doi: 10.3390/biomedicines13102460. PMID 41153743
- [Background] Serafin M, Maka M, Szostek J, Kania I, Jablonska B, Mrowiec S. Side-Specific Prognostic Factors in Colon Cancer: A Retrospective Analysis of Right- and Left-Sided Tumors. Cancers (Basel). 2025 Oct 14;17(20):3315. doi: 10.3390/cancers17203315. PMID 41154372
- [Background] Miranda J, Torri GB, Andreia Maria da Silva M, Monjardim G, Mariussi M, Schmitt LG, Wiethan CP, Ghezzi TL, Ghezzi CLA, Altmayer S, Dias AB, Horvat N. CT diagnostic performance for preoperative staging of colon cancer: a systematic review and meta-analysis. Eur Radiol. 2025 Aug 6. doi: 10.1007/s00330-025-11850-4. Online ahead of print. PMID 40767870
- [Background] Platt JR, Elliott F, Handley K, Magill L, Quirke P, Seymour MT, West NP, Morton D, Seligmann J, Tolan DJM. CT staging performance in an international trial of neoadjuvant chemotherapy for locally advanced colon cancer. Br J Radiol. 2025 Dec 1;98(1176):2175-2183. doi: 10.1093/bjr/tqaf217. PMID 40848246
- [Background] Gosavi R, Heriot A, Narasimhan V, Warrier SK. Perspectives of the Use of Neoadjuvant Therapy in the Management of Locally Advanced and Locally Recurrent Colon Cancer: A Bi-National Survey of Colorectal Surgeons. Asia Pac J Clin Oncol. 2025 Oct 13. doi: 10.1111/ajco.70035. Online ahead of print. PMID 41084117
- [Background] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089
- [Background] Patel RD, Patel B, Crnogorac-Jurcevic T. Extracellular Vesicle-Derived miRNAs as Diagnostic Biomarkers for Pancreatic Ductal Adenocarcinoma: A Systematic Review of Methodological Rigour and Clinical Applicability. Biomark Insights. 2025 Oct 25;20:11772719251381960. doi: 10.1177/11772719251381960. eCollection 2025. PMID 41180592
- [Background] Xia Y, Li B, Huang Z, Li X, Liu X, Zeng S, Fan Y, Yin J. Entropy-Driven Nucleic Acid Amplifier Based on Spatial Confinement as a "Booster" for Detection of Extracellular Vesicle MicroRNAs to Diagnose Gastric Cancer and Monitor Therapeutic Response. Anal Chem. 2025 Nov 25;97(46):25782-25796. doi: 10.1021/acs.analchem.5c05375. Epub 2025 Nov 3. PMID 41182092
- [Background] Yaghobinejad M, Naji M, Alizadeh AM, Aryanezhad S, Khalighfard S, Asadollahi P, Takzare N, Rastegar T. Identification and validation of stage-specific microRNAs and target genes for prostate cancer: Utilizing bioinformatics tools for diagnostic marker discovery. PLoS One. 2025 Nov 4;20(11):e0315366. doi: 10.1371/journal.pone.0315366. eCollection 2025. PMID 41187218